CLINICAL TRIAL: NCT01975246
Title: An Eight-week Randomised Double-blind Study to Compare the Efficacy and Safety of Telmisartan 80 mg and Amlodipine 5 mg and Hydrochlorothiazide 12.5 mg vs. Telmisartan 80 mg and Amlodipine 5 mg in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Telmisartan 80 mg and Amlodipine 5 mg
Brief Title: Add-on to Micamlo BP Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1348.1
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination; Hydrochlorothiazide

ARMS (2):
- Telmisartan+amlodipine+HCTZ (Experimental): telmisartan 80 mg + amlodipine 5 mg fixed dose combination (FDC) and hydrochlorothiazide (HCTZ) 12.5 mg tablet
  Interventions: Drug: Telmisartan + amlodipine; Drug: hydrochlorothiazide
- Telmisartan+amlodipine (Active Comparator): telmisartan 80 mg + amlodipine 5 mg fixed dose combination (FDC) and placebo matching hydrochlorothiazide 12.5 mg tablet
  Interventions: Drug: Telmisartan + amlodipine; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan + amlodipine — FDC tablet
  Arms: Telmisartan+amlodipine+HCTZ
Drug: hydrochlorothiazide — tablet
  Arms: Telmisartan+amlodipine+HCTZ
Drug: Telmisartan + amlodipine — FDC tablet
  Arms: Telmisartan+amlodipine
Drug: Placebo — placebo matching hydrochlorothiazide tablet
  Arms: Telmisartan+amlodipine

SUMMARY:
This is a multi-centre, randomised, double-blind, active-controlled, parallel-group comparative trial to compare the fixed dose combination (FDC) of telmisartan 80 mg +hydrochlorothiazide 12.5 mg and amlodipine 5 mg (T80/A5/H12.5 mg) to telmisartan 80 mg+ amlodipine 5 mg (T80/A5 mg) in blood pressure lowering effect at week 8, the end of the double-blind period in essential hypertensive patients who fail to respond adequately to telmisartan 80 mg+ amlodipine 5 mg. Patients are assigned to one of the two groups after a 6-week open-label run-in period taking T80/A5 mg.

ELIGIBILITY:
Inclusion criteria:

* Essential hypertensive patients who have already taking 2 or 3 antihypertensive drugs and mean seated diastolic blood pressure (DBP) must be >=90 and <=114 mmHg and mean seated systolic blood pressure (SBP) must be =<200 mmHg
* Able to stop all current antihypertensive drugs (other than study medication) from Visit 1b through the end of the trial without risk to the patient based on the investigator's opinion
* Age 20 years or older

Exclusion criteria:

* Patients with known or suspected secondary hypertension
* Patients with clinically relevant cardiac arrhythmia
* Congestive heart failure with New York Heart Association (NYHA) functional class III-IV
* Patients with recent cardiovascular events
* Patients with recent stroke events
* Patients with a history of sudden deterioration of renal function with angiotensin II receptor blockers or angiotensin converting enzyme inhibitors; or patients with post-renal transplant or post-nephrectomy
* Patients with hepatic and/or renal dysfunction
* Pre-menopausal women who are nursing or pregnant

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- Japan (30):
  - 1348.1.015 Boehringer Ingelheim Investigational Site, Atsubetsu-ku,Sapporo,Hokkaido
  - 1348.1.006 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 1348.1.002 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1348.1.005 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1348.1.031 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1348.1.030 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1348.1.033 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1348.1.016 Boehringer Ingelheim Investigational Site, Chuo-ku,Sapporo,Hokkaido
  - 1348.1.021 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1348.1.024 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1348.1.028 Boehringer Ingelheim Investigational Site, Itoshima, Fukuoka
  - 1348.1.027 Boehringer Ingelheim Investigational Site, Katsushika-ku, Tokyo
  - 1348.1.001 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 1348.1.009 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka
  - 1348.1.029 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka
  - 1348.1.014 Boehringer Ingelheim Investigational Site, Kiyose,Tokyo
  - 1348.1.003 Boehringer Ingelheim Investigational Site, Koto-ku, Tokyo
  - 1348.1.022 Boehringer Ingelheim Investigational Site, Mihama-ku, Chiba, Chiba
  - 1348.1.004 Boehringer Ingelheim Investigational Site, Miyagino-ku, Sendai, Miyagi
  - 1348.1.017 Boehringer Ingelheim Investigational Site, Moriya, Ibaraki
  - 1348.1.013 Boehringer Ingelheim Investigational Site, Naka-ku,Yokohama,Kanagawa
  - 1348.1.018 Boehringer Ingelheim Investigational Site, Nishi-ku, Fukuoka, Fukuoka
  - 1348.1.007 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1348.1.020 Boehringer Ingelheim Investigational Site, Sakaide, Kagawa
  - 1348.1.025 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1348.1.026 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1348.1.008 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1348.1.032 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1348.1.019 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1348.1.023 Boehringer Ingelheim Investigational Site, Toshima-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is randomised, double-blind, active-control, parallel-group comparison
Groups:
- Telmisartan and Amlodipine+HCTZ: Subjects who were orally administered once daily with fixed dose combination (FDC) tablet of telmisartan 80 mg and amlodipine 5 mg+ hydrochlorothiazide (HCTZ) 12.5 mg tablet.
- Telmisartan+Amlodipine: Subjects who were orally administered once daily with the fixed-dose combination tablet of telmisartan 80 mg and amlodipine 5 mg + placebo matching to hydrochlorothiazide 12.5 mg tablet
Period: Overall Study
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine
Started | 149 | 160
Completed | 145 | 158
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other than stated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set consisted of all patients who were randomised to the double-blind period and took at least 1 dose of the randomised treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine | Total
Number analyzed (Participants) | 149 | 160 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (9.1) | 55.0 (9.7) | 54.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 127 | 130 | 257

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated DBP at Trough After 8 Weeks of the Double-blind Period.
Description: Change from baseline in mean seated diastolic blood pressure (DBP) at trough after 8 weeks of the double-blind period. After patients had rested in a seated position for approximately 5 minutes, blood pressure was measured 3 times at approximately 2-minute intervals. The mean of the 3 measurements are used as endpoints.
Time Frame: baseline and week 8
Population: Full analysis set (FAS): This analysis set was, conforming to the intent-to-treat principle, defined as all patients i) included in the treated set; and ii) taking measurements of seated DBP at reference baseline and at 1 or more time points during the double-blind period.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine
Number analyzed (Participants) | 147 | 160
mmHg | -8.4 (0.5) | -4.5 (0.5)
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine+HCTZ vs Telmisartan+Amlodipine; The last observation carried forward (LOCF) method was applied for missing data, where the value from the measurements at the closest preceding visit replaced the missing value; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes baseline DBP as a linear covariate, and treatment and center as fixed effects; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-5.3 to -2.4], Standard Error of Mean 0.7

2. Secondary Outcome: Change From Baseline in Mean Seated SBP at Trough After 8 Weeks of the Double-blind Period.
Description: Change from baseline in mean seated systolic blood pressure (SBP) at trough after 8 weeks of the double-blind period. After patients had rested in a seated position for approximately 5 minutes, blood pressure was measured 3 times at approximately 2-minute intervals. The mean of the 3 measurements are used as endpoints.
Time Frame: baseline and week 8
Population: FAS
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine
Number analyzed (Participants) | 147 | 160
mmHg | -12.3 (0.8) | -6.9 (0.8)
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine+HCTZ vs Telmisartan+Amlodipine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Model includes baseline SBP as a linear covariate, and treatment and center as fixed effects; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-7.6 to -3.1], Standard Error of Mean 1.1

3. Secondary Outcome: The Proportion of Patients With DBP<90 mmHg and SBP<140 mmHg as Seated Blood Pressure at Trough After 8 Weeks of the Double-blind Period
Description: Patients with trough seated DBP =>90 mmHg or trough seated SBP >=140 mmHg at baseline were analysed.
Time Frame: baseline and week 8
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine
Number analyzed (Participants) | 147 | 160
percentage of participants | 51.7 [43.3 to 60.0] | 36.9 [29.4 to 44.9]
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine+HCTZ vs Telmisartan+Amlodipine; The Non-completers considered failure (NCF) method was applied for missing data, where missing data due to early discontinuation will be replaced as "failure" up to the planned final visit to be reached by all patients; Test type: Superiority or Other; p < 0.0051, Regression, Logistic; Logistic regression model includes treatment and center as fixed effects; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.2 to 3.4]

ADVERSE EVENTS:
Time Frame: From first drug administration until 24 hours after the last drug administration, up to 71 days.
Arm/Group | Telmisartan and Amlodipine+HCTZ | Telmisartan+Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/160
Other Adverse Events (participants affected / at risk) | 36/149 | 14/160
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan and Amlodipine+HCTZ (N=149) | Telmisartan+Amlodipine (N=160)
Nasopharyngitis (Infections and infestations) | 9 | 9
Blood uric acid increased (Investigations) | 20 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.